CLINICAL TRIAL: NCT05383365
Title: The Effectiveness of Deep Neck Flexor Exercises in Comparison With Myofascial Release of Suboccipital Muscle on Pain and Forward Head Posture in People With Chronic Tension-type Headache and Forward Head Posture
Brief Title: Deep Neck Flexor Exercises Versus Myofascial Release of Suboccipital Muscles in Chronic Tension-type Headache
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Iran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IR.IUMS.REC.1400.1239
Record Dates: First submitted 2022-04-21; First posted 2022-05-20 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-02

CONDITIONS: Chronic Tension-Type Headache
Keywords: Chronic tension-type headache; Chronic primary headache; Forward head posture; Deep neck flexor exercise; Pressure biofeedback; Myofascial release; Pressure pain threshold; Quality of life; Disability

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suboccipital Myofascial Release (Experimental): The therapist places the supinated forearm on the bed and positions the tips of the middle three fingers inferior to the occiput bone and the head is supported by the thenar eminences
  Interventions: Other: Suboccipital Myofascial Release(MFR) with sham Deep Neck Flexor(DNF)exercise
- Deep Neck Flexor Exercise (Experimental): After placing the airbag of PBU under the occiput bone in the supine position and inflating it to a base pressure of 11 mmHg, the participant will increase the pressure to 12 mmHg by nodding action.
  Interventions: Other: Deep Neck Flexor(DNF)exercise with sham Suboccipital Myofascial Release(MFR)

INTERVENTIONS:
Other: Suboccipital Myofascial Release(MFR) with sham Deep Neck Flexor(DNF)exercise — The treatment includes Suboccipital MFR in the supine position.The therapist places the supinated forearm on the bed and positions the tips of the middle three fingers inferior to the occiput bone and the head is supported by the thenar eminences.The therapist will develop a line of tension through the suboccipital tissues by supinating the forearms and pulling apart two hands from each other;Then, for the second level in the first position of hands,pressure is applied to the anterior and superior direction.The pressure is held and increased until the therapist feels the decrease of muscle tone.These techniques last 10 minutes.
  Another intervention in this group is the sham DNF exercise with a Pressure Biofeedback Unit(PBU).Considering that minimum detective change with PBU is 15 mmHg; After placing the airbag of PBU under the occiput bone in the supine position and inflating it to a base pressure of 11 mmHg,the participant will increase the pressure to 12 mmHg by nodding action.
  Arms: Suboccipital Myofascial Release
Other: Deep Neck Flexor(DNF)exercise with sham Suboccipital Myofascial Release(MFR) — The treatments include the DNF exercise with a PBU. The treatment is performed in the supine position and the airbag is placed under the occiput bone and is inflated to a base pressure of 20 mmHg. The participant will increase and hold the pressure to a special point by nodding action. The exercise is repeated for 3 sets, in each set 2 mm Hg is added to the pressure. The pressure will be increased from 22 to 32 mm Hg during 4-week of treatment, and each goal is held for 10 seconds and repeated 10 times. There will be 5 sec of rest between each repetition and 2 min of rest between each set.
  Another intervention in this group is sham MFR. The therapist's hands will be placed only inferior to the occipital bone and a superficial touch is applied without any upward or lateral pressure. sham treatment in this group, like the opposite group, lasts 10 minutes.
  Arms: Deep Neck Flexor Exercise

SUMMARY:
According to the study of the burden of diseases in 2018, tension-type headache(TTH) is the most common type of primary headache and ranks third in terms of prevalence among 328 diseases and injuries in 195 countries from 1990 to 2016. Suffering from this disorder (especially chronic type) reduces the quality of life of patients.

The main objective of this study is to compare the effects of myofascial release of suboccipital muscles as a bottom-up intervention and Deep Neck Flexor(DNF) exercises with Pressure Biofeedback Unit(PBU) as a top-down intervention on headache parameters, the intensity of Forward Head Posture(FHP), disability, quality of life, and suboccipital Pressure Pain Threshold(PPT) in patients with chronic tension-type headache with forward head posture.

DETAILED DESCRIPTION:
Previous studies demonstrated that suboccipital active Trigger Points(TrPs) and forward head posture were associated with Chronic Tension-Type Headache(CTTH) and they can aggravate parameters of headache in these patients. The greater suboccipital muscle contraction, as would be exexpected in greater FHP, the more the nociceptive input into the trigeminal nucleus caudalis, and the lower the headache or pain threshold, consistent with increased central sensitization; Therefore it is important to evaluate the effectiveness of interventions on FHP and suboccipital active TrPs in patients with CTTH.

The main objective of this study is to compare the effects of myofascial release of suboccipital muscles as a bottom-up intervention and deep neck flexor exercises with a pressure biofeedback unit as a top-down intervention.

Primary outcomes will be the intensity of headache and FHP. headache duration and frequency, disability, quality of life, and pain pressure threshold will be considered as secondary outcomes.

In this study, a double-dummy randomized clinical trial, 44 participants will be divided into two groups of DNF exercises with pressure biofeedback combined with sham MFR (first group) and sub-occipital MFR combined with sham DNF exercises(second group). The intervention will take place over a 4-week period, with three 1-hour sessions a week, totaling 12 treatment sessions. this study has a 6-week follow-up.

This study is a double-blind study in which the participants, the person evaluating the outcome, and the statistician of the data will be blinded to the allocation of patients to the two treatment groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 55 years;
2. based on ICHD-3, Headache that occurs 15 days per month and lasts on average for >3 months (180 days per year), lasting hours to days, or unremitting, and has at least two of the following four characteristics recognized as CTTH: bilateral location, pressing or tightening (non-pulsating) quality, mild or moderate intensity, not aggravated by routine physical activity such as walking or climbing stairs and both of the following: no more than one of photophobia, phonophobia or mild nausea, neither moderate or severe nausea nor vomiting;
3. Dosage and type of prophylactic medication have not changed in the months before the beginning of the trial;
4. The participant does not intend to change the dosage and type of prophylactic medication during the study;
5. CVA less than 49 degrees,
6. Participants have the ability to understand and read Persian to complete the questionnaire.

Exclusion Criteria:

1. Participants with infrequent ETTH, or other primary or secondary types of headache;
2. Pain aggravated by movement of the head;
3. Severe pain or significant decrease in ROM of the cervical spine;
4. Previous trauma to the cervical spine;
5. History of injection, surgery, severe disc protrusion, or neck or shoulder fracture that affects treatment;
6. Metabolic or Neurological disorders such as Bow hunter's syndrome or epilepsy;
7. Taking more than 200 pieces of morphine or other strong analgesics per month;
8. Physiotherapy treatment for headache within 6 months before starting treatment;
9. Joint stiffness, atherosclerosis, or advanced osteoarthritis;
10. Manual contraindication includes: (a)The participant has substance or alcohol abuse; (b)For whatever reason, the participant does not want to be touched by the therapist; (c)Symptoms are severe and irritating; (d)Underlying diseases (such as rheumatoid arthritis) or metabolic disorders (such as osteoporosis or soft tissue laxity of the treatment area);
11. Pregnancy;
12. Spielberger State-Trait Anxiety Inventory (STAI) scores more than 85;
13. Absence of two consecutive sessions and more than treatment sessions.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Intensity of headache using by Numeric Pain Rating Scale(NPRS) | Change in the intensity of headache after the end of 12 treatment sessions compared to baseline and change from Baseline at 6-week follow up
  In the initial evaluation of the participants, the pain intensity will be determined based on the NPRS on a scale of 0-100. For this purpose, the participant is asked to mark their average pain intensity in the last month on a 100 cm line without scaling from zero to 100. The number zero indicates the absence of pain and the number 100 indicates the most pain the person has experienced in their life. The marked point is then measured with a ruler. Participants are asked to record their average intensity of pain during the past month on the Headache Questionnaire.
  Evaluation of the headache intensity will be done after treatment and in a 6 weeks follow-up by the headache diary; For this purpose, during the four weeks of treatment and up to 6 weeks after the treatment, the participant is asked to record the amount of headache intensity on a daily basis in this diary.
intensity of Forward Head Posture(FHP) using by Craniovertebral Angle(CVA) | Change in the intensity of Forward Head Posture after the end of 12 treatment sessions compared to baseline and change from Baseline at 6-week follow up
  The amount of is measured using the photogrammetric method of body profile for measuring the FHP. This method has high reliability (ICC = 0.83). This angle will be assessed in sitting posture from profile view, in this picture the spinous process of the seventh cervical vertebra and tragus of the ear is marked with landmarks. Photography is done with a camera (smartphone iPhone 13 pro, Apple Inc) with a magnification of 1 and is placed at a certain distance from the person on a fixed base. Finally, the images are transferred to a computer and the angle between the line connecting the ear tragus to the spinous process of the seventh cervical vertebra and the horizon line is measured using Kinovea software (ICC=.99).

SECONDARY OUTCOMES:
Duration of headache using by headache questionnaire and diary | Change in the duration of headache after the end of 12 treatment sessions compared to baseline and change from Baseline at 6-week follow up
  The duration of pain will be determined based on the average number of hours a person experiences a headache in a month. Participants are asked to record their average duration of pain during the past month on the Headache Questionnaire.
  Evaluation of the headache duration will be done after treatment and in a 6-week follow-up by the headache diary; For this purpose, during the four weeks of treatment and up to 6 weeks after the treatment, the participant is asked to record the amount of headache duration on a daily basis in this diary.
Frequency of headache using by headache questionnaire and diary | Change in the frequency of headache after the end of 12 treatment sessions compared to baseline and change from Baseline at 6-week follow up
  The frequency of headaches is based on the number of days in the month that the person experiences the headache. Participants are asked to record their average frequency of pain during the past month on the Headache Questionnaire.
  Evaluation of the headache frequency will be done after treatment and in a 6 week follow-up by the headache diary; For this purpose, during the four weeks of the treatment and up to 6 weeks after treatment, the participant is asked to record the amount of headache frequency on a daily basis in this diary.
Disability using by Henry Ford Hospital Headache Disability Inventory (HDI) questionnaire | Change in the disability after the end of 12 treatment sessions compared to baseline and change from Baseline at 6-week follow up
  The Persian version of the Henry Ford Hospital Headache Disability Inventory (HDI) questionnaire will be used to assess the amount of disability. The questionnaire has 25 questions that include functional and emotional subsets, and each "yes" answer is a 4-point answer, each "sometimes" answer is a 2-point answer, and each "no" answer is a zero-point answer. This questionnaire consists of 12 questions in the functional field with a maximum score of 48 and 13 questions in the emotional field with a maximum score of 52, which adds up to 100 points. The higher the score, the greater the disability due to the headache. If, as a result of the therapeutic approach, a score equal to or greater than 29 points is seen in this questionnaire, it indicates significant changes. The internal consistency of the Persian version of this questionnaire with Cronbach's alpha is 0.91 for the whole questionnaire, 0.82 for the functional area and 0.86 for the emotional area (ICC = 0.97).
Quality of life using by Headache Impact Test -6 (HIT-6) questionnaire | Change in the quality of life after the end of 12 treatment sessions compared to baseline and change from Baseline at 6-week follow up
  The Persian version of the Headache Impact Test -6 (HIT-6) questionnaire will be used. This short questionnaire includes 6 questions that are a reminder of the last 4 weeks. Scores are between 36 and 78, and higher scores indicate a higher intensity of headache and a greater impact of headache on a person's quality of life. This questionnaire is used to measure the effect of headache and its treatment on a person's functional status and quality of life, and its psychological characteristics have been extensively studied. The questions in this questionnaire cover problems including pain, ability to perform daily life activities, social functioning, energy/fatigue, cognitive function, and psychological problems. The reliability coefficient of this questionnaire in different researches through retesting, peer forms, and internal stability are 0.8, 0.9, and 0.89, respectively.
Pressure Pain Threshold(PPT) using by algometer | Change in the pain pressure threshold after the end of 12 treatment sessions compared to baseline and change from Baseline at 6-week follow up
  An algometer (JTECH Medical, made in the USA) is used to assess the pain pressure threshold of suboccipital muscles. In this method, the participant is lying on a Manual Physical Therapy Table (MPT) with a cavity for placing the face lying down and an algometer with a 1 cm^2 cross-sectional area vertically and at a speed of about 1 kg / cm^2 at the bottom of the occiput bone and outside of the upper trapezius muscle are placed on both sides. Pressure is applied until the feeling of pressure turns into a feeling of pain and the participant is asked to announce the moment of onset of pain. The measurement is repeated 3 times with an interval of 30 seconds, then the average is calculated. It should be noted that this device has high reliability (ICC = 0.78 - 0.93)

CONTACTS AND LOCATIONS:
Overall Officials: Mobina Ahmadi, MSc student, Principal Investigator — MSc student; Mohammadreza Pourahmadi, Study Director — Professor Assisstant

IPD SHARING:
Plan to Share IPD: Yes
The data sets of this study will be available on a reasonable request to the corresponding author
Supporting Information: Study Protocol
Time Frame: starting 6 months after the publication
Access Criteria: The data will be available for physical therapists working in academic institutions and also clinicians working in the field of musculoskeletal disorders and headaches. The raw data and results of this study can be used in future relevant systematic reviews. Thus, the raw data and results of this study will be available for researchers working in the field of tension-type headache. Applicants can contact Mobina Ahmadi by Email.
  Email Address:M.oahmadi@ymail.com Applicants should explain their project and how the data/documents of the study will be used in their project in detail. Then, the data/documents files will be sent by email to applicants on request. This process may take 10-12 working days.

REFERENCES:
- [Background] Steiner TJ, Stovner LJ, Jensen R, Uluduz D, Katsarava Z; Lifting The Burden: the Global Campaign against Headache. Migraine remains second among the world's causes of disability, and first among young women: findings from GBD2019. J Headache Pain. 2020 Dec 2;21(1):137. doi: 10.1186/s10194-020-01208-0. No abstract available. PMID 33267788
- [Background] Headache Classification Committee of the International Headache Society (IHS). The International Classification of Headache Disorders, 3rd edition (beta version). Cephalalgia. 2013 Jul;33(9):629-808. doi: 10.1177/0333102413485658. No abstract available. PMID 23771276
- [Background] Stovner Lj, Hagen K, Jensen R, Katsarava Z, Lipton R, Scher A, Steiner T, Zwart JA. The global burden of headache: a documentation of headache prevalence and disability worldwide. Cephalalgia. 2007 Mar;27(3):193-210. doi: 10.1111/j.1468-2982.2007.01288.x. PMID 17381554
- [Background] GBD 2016 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 328 diseases and injuries for 195 countries, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet. 2017 Sep 16;390(10100):1211-1259. doi: 10.1016/S0140-6736(17)32154-2. PMID 28919117
- [Background] Ashina S, Buse DC, Bjorner JB, Bendtsen L, Lyngberg AC, Jensen RH, Lipton RB. Health-related quality of life in tension-type headache: a population-based study. Scand J Pain. 2021 Jan 25;21(4):778-787. doi: 10.1515/sjpain-2020-0166. Print 2021 Oct 26. PMID 33544560
- [Background] GBD 2016 Headache Collaborators. Global, regional, and national burden of migraine and tension-type headache, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet Neurol. 2018 Nov;17(11):954-976. doi: 10.1016/S1474-4422(18)30322-3. PMID 30353868
- [Background] Fumal A, Schoenen J. Tension-type headache: current research and clinical management. Lancet Neurol. 2008 Jan;7(1):70-83. doi: 10.1016/S1474-4422(07)70325-3. PMID 18093564
- [Background] Bendtsen L. Central sensitization in tension-type headache--possible pathophysiological mechanisms. Cephalalgia. 2000 Jun;20(5):486-508. doi: 10.1046/j.1468-2982.2000.00070.x. PMID 11037746
- [Background] Fernandez-de-las-Penas C, Cuadrado ML, Arendt-Nielsen L, Simons DG, Pareja JA. Myofascial trigger points and sensitization: an updated pain model for tension-type headache. Cephalalgia. 2007 May;27(5):383-93. doi: 10.1111/j.1468-2982.2007.01295.x. Epub 2007 Mar 14. PMID 17359516
- [Background] Rasmussen BK. Migraine and tension-type headache in a general population: precipitating factors, female hormones, sleep pattern and relation to lifestyle. Pain. 1993 Apr;53(1):65-72. doi: 10.1016/0304-3959(93)90057-V. PMID 8316392
- [Background] Wober C, Holzhammer J, Zeitlhofer J, Wessely P, Wober-Bingol C. Trigger factors of migraine and tension-type headache: experience and knowledge of the patients. J Headache Pain. 2006 Sep;7(4):188-95. doi: 10.1007/s10194-006-0305-3. Epub 2006 Aug 11. PMID 16897622
- [Background] Marcus DA, Scharff L, Mercer S, Turk DC. Musculoskeletal abnormalities in chronic headache: a controlled comparison of headache diagnostic groups. Headache. 1999 Jan;39(1):21-7. doi: 10.1046/j.1526-4610.1999.3901021.x. PMID 15613190
- [Background] Griegel-Morris P, Larson K, Mueller-Klaus K, Oatis CA. Incidence of common postural abnormalities in the cervical, shoulder, and thoracic regions and their association with pain in two age groups of healthy subjects. Phys Ther. 1992 Jun;72(6):425-31. doi: 10.1093/ptj/72.6.425. PMID 1589462
- [Background] Chu ECP, Lo FS, Bhaumik A. Plausible impact of forward head posture on upper cervical spine stability. J Family Med Prim Care. 2020 May 31;9(5):2517-2520. doi: 10.4103/jfmpc.jfmpc_95_20. eCollection 2020 May. PMID 32754534
- [Background] Fernandez-de-las-Penas C, Alonso-Blanco C, Cuadrado ML, Pareja JA. Forward head posture and neck mobility in chronic tension-type headache: a blinded, controlled study. Cephalalgia. 2006 Mar;26(3):314-9. doi: 10.1111/j.1468-2982.2005.01042.x. PMID 16472338
- [Background] Fernandez-de-las-Penas C, Alonso-Blanco C, Cuadrado ML, Gerwin RD, Pareja JA. Trigger points in the suboccipital muscles and forward head posture in tension-type headache. Headache. 2006 Mar;46(3):454-60. doi: 10.1111/j.1526-4610.2006.00288.x. PMID 16618263
- [Background] Fernandez-de-las-Penas C, Alonso-Blanco C, Cuadrado ML, Pareja JA. Neck mobility and forward head posture are not related to headache parameters in chronic tension-type headache. Cephalalgia. 2007 Feb;27(2):158-64. doi: 10.1111/j.1468-2982.2006.01247.x. PMID 17257237
- [Background] Torelli P, Jensen R, Olesen J. Physiotherapy for tension-type headache: a controlled study. Cephalalgia. 2004 Jan;24(1):29-36. doi: 10.1111/j.1468-2982.2004.00633.x. PMID 14687010
- [Background] Fernández-de-las-Peñas C, Arendt-Nielsen L, Gerwin RD. Tension-type and cervicogenic headache: pathophysiology, diagnosis, and management: Jones & Bartlett Publishers; 2010.
- [Background] Fernandez-de-Las-Penas C, Florencio LL, Plaza-Manzano G, Arias-Buria JL. Clinical Reasoning Behind Non-Pharmacological Interventions for the Management of Headaches: A Narrative Literature Review. Int J Environ Res Public Health. 2020 Jun 9;17(11):4126. doi: 10.3390/ijerph17114126. PMID 32527071
- [Background] Lai AKM, Arnold AS, Wakeling JM. Why are Antagonist Muscles Co-activated in My Simulation? A Musculoskeletal Model for Analysing Human Locomotor Tasks. Ann Biomed Eng. 2017 Dec;45(12):2762-2774. doi: 10.1007/s10439-017-1920-7. Epub 2017 Sep 12. PMID 28900782
- [Background] Castien R, Blankenstein A, van der Windt D, Heymans MW, Dekker J. The working mechanism of manual therapy in participants with chronic tension-type headache. J Orthop Sports Phys Ther. 2013 Oct;43(10):693-9. doi: 10.2519/jospt.2013.4868. Epub 2013 Sep 9. PMID 24256171
- [Background] Lee E, Lee S. Impact of Cervical Sensory Feedback for Forward Head Posture on Headache Severity and Physiological Factors in Patients with Tension-type Headache: A Randomized, Single-Blind, Controlled Trial. Med Sci Monit. 2019 Dec 15;25:9572-9584. doi: 10.12659/MSM.918595. PMID 31838486
- [Background] Cosio D, Lin E. Role of Active Versus Passive Complementary and Integrative Health Approaches in Pain Management. Glob Adv Health Med. 2018 Apr 10;7:2164956118768492. doi: 10.1177/2164956118768492. eCollection 2018. PMID 29662720
- [Background] Cho SH. The effect of suboccipital muscle inhibition and posture correction exercises on chronic tension-type headaches. J Back Musculoskelet Rehabil. 2021;34(6):989-996. doi: 10.3233/BMR-191667. PMID 33935056
- [Background] Choi W. Effect of 4 Weeks of Cervical Deep Muscle Flexion Exercise on Headache and Sleep Disorder in Patients with Tension Headache and Forward Head Posture. Int J Environ Res Public Health. 2021 Mar 25;18(7):3410. doi: 10.3390/ijerph18073410. PMID 33806089
- [Background] Victoria Espi-Lopez G, Arnal-Gomez A, Arbos-Berenguer T, Gonzalez AAL, Vicente-Herrero T. Effectiveness of Physical Therapy in Patients with Tension-type Headache: Literature Review. J Jpn Phys Ther Assoc. 2014;17(1):31-38. doi: 10.1298/jjpta.Vol17_005. PMID 25792906
- [Background] Elizagaray-Garcia I, Beltran-Alacreu H, Angulo-Diaz S, Garrigos-Pedron M, Gil-Martinez A. Chronic Primary Headache Subjects Have Greater Forward Head Posture than Asymptomatic and Episodic Primary Headache Sufferers: Systematic Review and Meta-analysis. Pain Med. 2020 Oct 1;21(10):2465-2480. doi: 10.1093/pm/pnaa235. PMID 33118601
- [Background] Jull G, Trott P, Potter H, Zito G, Niere K, Shirley D, Emberson J, Marschner I, Richardson C. A randomized controlled trial of exercise and manipulative therapy for cervicogenic headache. Spine (Phila Pa 1976). 2002 Sep 1;27(17):1835-43; discussion 1843. doi: 10.1097/00007632-200209010-00004. PMID 12221344
- [Background] Jull GA, Falla D, Vicenzino B, Hodges PW. The effect of therapeutic exercise on activation of the deep cervical flexor muscles in people with chronic neck pain. Man Ther. 2009 Dec;14(6):696-701. doi: 10.1016/j.math.2009.05.004. Epub 2009 Jul 25. PMID 19632880
- [Background] Alghadir AH, Iqbal ZA. Effect of Deep Cervical Flexor Muscle Training Using Pressure Biofeedback on Pain and Forward Head Posture in School Teachers with Neck Pain: An Observational Study. Biomed Res Int. 2021 May 22;2021:5588580. doi: 10.1155/2021/5588580. eCollection 2021. PMID 34095302
- [Background] Liang Z, Galea O, Thomas L, Jull G, Treleaven J. Cervical musculoskeletal impairments in migraine and tension type headache: A systematic review and meta-analysis. Musculoskelet Sci Pract. 2019 Jul;42:67-83. doi: 10.1016/j.msksp.2019.04.007. Epub 2019 Apr 25. PMID 31054485
- [Background] Kalmanson OA, Khayatzadeh S, Germanwala A, Scott-Young M, Havey RM, Voronov LI, Patwardhan AG. Anatomic considerations in headaches associated with cervical sagittal imbalance: A cadaveric biomechanical study. J Clin Neurosci. 2019 Jul;65:140-144. doi: 10.1016/j.jocn.2019.02.003. Epub 2019 Mar 12. PMID 30876933
- [Background] Falsiroli Maistrello L, Geri T, Gianola S, Zaninetti M, Testa M. Effectiveness of Trigger Point Manual Treatment on the Frequency, Intensity, and Duration of Attacks in Primary Headaches: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Front Neurol. 2018 Apr 24;9:254. doi: 10.3389/fneur.2018.00254. eCollection 2018. PMID 29740386
- [Background] Falsiroli Maistrello L, Rafanelli M, Turolla A. Manual Therapy and Quality of Life in People with Headache: Systematic Review and Meta-analysis of Randomized Controlled Trials. Curr Pain Headache Rep. 2019 Aug 10;23(10):78. doi: 10.1007/s11916-019-0815-8. PMID 31401702
- [Background] Kamonseki DH, Lopes EP, van der Meer HA, Calixtre LB. Effectiveness of manual therapy in patients with tension-type headache. A systematic review and meta-analysis. Disabil Rehabil. 2022 May;44(10):1780-1789. doi: 10.1080/09638288.2020.1813817. Epub 2020 Sep 12. PMID 32924640
- [Background] Ajimsha MS, Al-Mudahka NR, Al-Madzhar JA. Effectiveness of myofascial release: systematic review of randomized controlled trials. J Bodyw Mov Ther. 2015 Jan;19(1):102-12. doi: 10.1016/j.jbmt.2014.06.001. Epub 2014 Jun 13. PMID 25603749
- [Background] Williams ACC, Craig KD. Updating the definition of pain. Pain. 2016 Nov;157(11):2420-2423. doi: 10.1097/j.pain.0000000000000613. No abstract available. PMID 27200490
- [Background] Kendall FP ME, Provance PJG, Rodgers MM, Romani, RA ea. Muscles testing and function with posture and pain. Fifth ed2005.
- [Background] Neumann D. Kinesiology of the Musculoskeletal System - Foundations for Rehabilitation. Kinesiology of the Musculoskeletal System ed: elsevier; 2016.
- [Background] Lutz BJ, Bowers BJ. Understanding how disability is defined and conceptualized in the literature. Rehabil Nurs. 2003 May-Jun;28(3):74-8. doi: 10.1002/j.2048-7940.2003.tb02037.x. PMID 12747245
- [Background] Jabbari S, Salahzadeh Z, Sarbakhsh P, Rezaei M, Farhoudi M, Ghodrati M. Validity and Reliability of Persian Version of Henry Ford Hospital Headache Disability Inventory Questionnaire. Arch Iran Med. 2021 Oct 1;24(10):752-758. doi: 10.34172/aim.2021.111. PMID 34816697
- [Background] Haraldstad K, Wahl A, Andenaes R, Andersen JR, Andersen MH, Beisland E, Borge CR, Engebretsen E, Eisemann M, Halvorsrud L, Hanssen TA, Haugstvedt A, Haugland T, Johansen VA, Larsen MH, Lovereide L, Loyland B, Kvarme LG, Moons P, Norekval TM, Ribu L, Rohde GE, Urstad KH, Helseth S; LIVSFORSK network. A systematic review of quality of life research in medicine and health sciences. Qual Life Res. 2019 Oct;28(10):2641-2650. doi: 10.1007/s11136-019-02214-9. Epub 2019 Jun 11. PMID 31187410
- [Background] Zandifar A, Banihashemi M, Haghdoost F, Masjedi SS, Manouchehri N, Asgari F, Najafi MR, Ghorbani A, Zandifar S, Saadatnia M, White MK. Reliability and Validity of the Persian HIT-6 Questionnaire in Migraine and Tension-type Headache. Pain Pract. 2014 Sep;14(7):625-31. doi: 10.1111/papr.12120. Epub 2013 Nov 18. PMID 24237583
- [Background] Ylinen J. Pressure algometry. Aust J Physiother. 2007;53(3):207. doi: 10.1016/s0004-9514(07)70032-6. No abstract available. PMID 17899675
- [Background] Espi-Lopez GV, Gomez-Conesa A, Gomez AA, Martinez JB, Pascual-Vaca AO, Blanco CR. Treatment of tension-type headache with articulatory and suboccipital soft tissue therapy: A double-blind, randomized, placebo-controlled clinical trial. J Bodyw Mov Ther. 2014 Oct;18(4):576-85. doi: 10.1016/j.jbmt.2014.01.001. Epub 2014 Jan 10. PMID 25440210
- [Background] Bendtsen L, Bigal ME, Cerbo R, Diener HC, Holroyd K, Lampl C, Mitsikostas DD, Steiner TJ, Tfelt-Hansen P; International Headache Society Clinical Trials Subcommittee. Guidelines for controlled trials of drugs in tension-type headache: second edition. Cephalalgia. 2010 Jan;30(1):1-16. doi: 10.1111/j.1468-2982.2009.01948.x. PMID 19614696
- [Background] Berggreen S, Wiik E, Lund H. Treatment of myofascial trigger points in female patients with chronic tension-type headache - a randomized controlled trial. Advances in Physiotherapy. 2012;14(1):10-7.
- [Background] Kamali F, Mohamadi M, Fakheri L, Mohammadnejad F. Dry needling versus friction massage to treat tension type headache: A randomized clinical trial. J Bodyw Mov Ther. 2019 Jan;23(1):89-93. doi: 10.1016/j.jbmt.2018.01.009. Epub 2018 Jan 31. PMID 30691768
- [Background] Alvarez-Melcon AC, Valero-Alcaide R, Atin-Arratibel MA, Melcon-Alvarez A, Beneit-Montesinos JV. Effects of physical therapy and relaxation techniques on the parameters of pain in university students with tension-type headache: A randomised controlled clinical trial. Neurologia (Engl Ed). 2018 May;33(4):233-243. doi: 10.1016/j.nrl.2016.06.008. Epub 2016 Aug 1. English, Spanish. PMID 27491303
- [Background] DeStefano LAGPE. Greenman's principles of manual medicine. Philadelphia, Pa.; London: Lippincott Williams & Wilkins; 2010.
- [Background] Maitland GDMGD. Maitland's vertebral manipulation. Oxford; Boston: Butterworth-Heinemann; 2001.
- [Background] Youssef A. Photogrammetric Quantification of Forward Head Posture is Side Dependent in Healthy Participants and Patients with Mechanical Neck Pain. International Journal of Physiotherapy. 2016;3.
- [Background] Puig-Divi A, Escalona-Marfil C, Padulles-Riu JM, Busquets A, Padulles-Chando X, Marcos-Ruiz D. Validity and reliability of the Kinovea program in obtaining angles and distances using coordinates in 4 perspectives. PLoS One. 2019 Jun 5;14(6):e0216448. doi: 10.1371/journal.pone.0216448. eCollection 2019. PMID 31166989
- [Background] Lundqvist C, Benth JS, Grande RB, Aaseth K, Russell MB. A vertical VAS is a valid instrument for monitoring headache pain intensity. Cephalalgia. 2009 Oct;29(10):1034-41. doi: 10.1111/j.1468-2982.2008.01833.x. Epub 2009 Mar 12. PMID 19735531
- [Background] Jacobson GP, Ramadan NM, Aggarwal SK, Newman CW. The Henry Ford Hospital Headache Disability Inventory (HDI). Neurology. 1994 May;44(5):837-42. doi: 10.1212/wnl.44.5.837. PMID 8190284
- [Background] Florencio LL, Giantomassi MC, Carvalho GF, Goncalves MC, Dach F, Fernandez-de-Las-Penas C, Bevilaqua-Grossi D. Generalized Pressure Pain Hypersensitivity in the Cervical Muscles in Women with Migraine. Pain Med. 2015 Aug;16(8):1629-34. doi: 10.1111/pme.12767. Epub 2015 Apr 30. PMID 25929269
- [Background] Ylinen J, Nykanen M, Kautiainen H, Hakkinen A. Evaluation of repeatability of pressure algometry on the neck muscles for clinical use. Man Ther. 2007 May;12(2):192-7. doi: 10.1016/j.math.2006.06.010. Epub 2006 Sep 7. PMID 16956783
- [Background] Garrett TR, Youdas JW, Madson TJ. Reliability of measuring forward head posture in a clinical setting. J Orthop Sports Phys Ther. 1993 Mar;17(3):155-60. doi: 10.2519/jospt.1993.17.3.155. PMID 8472080
- [Background] Jeong ED, Kim CY, Kim SM, Lee SJ, Kim HD. Short-term effects of the suboccipital muscle inhibition technique and cranio-cervical flexion exercise on hamstring flexibility, cranio-vertebral angle, and range of motion of the cervical spine in subjects with neck pain: A randomized controlled trial. J Back Musculoskelet Rehabil. 2018;31(6):1025-1034. doi: 10.3233/BMR-171016. PMID 30248030
- [Background] Stanborough M. Direct Release Myofascial Technique-An Illustrated Guide for Practitioners. first ed: elsevier; 2004.
- [Background] Faustino D, Vieira A, Candotti CT, Detogni Schmit EF, Rios Xavier MF, Lunelli VA, Loss JF. Repeatability and reproducibility of the pressure biofeedback unit. J Bodyw Mov Ther. 2021 Jul;27:560-564. doi: 10.1016/j.jbmt.2021.04.017. Epub 2021 Apr 28. PMID 34391287
- [Background] Rezaeian T, Mosallanezhad Z, Nourbakhsh MR, Ahmadi M, Nourozi M. The Impact of Soft Tissue Techniques in the Management of Migraine Headache: A Randomized Controlled Trial. J Chiropr Med. 2019 Dec;18(4):243-252. doi: 10.1016/j.jcm.2019.12.001. Epub 2020 Aug 1. PMID 32952469
- [Background] Pryse-Phillips W, Findlay H, Tugwell P, Edmeads J, Murray TJ, Nelson RF. A Canadian population survey on the clinical, epidemiologic and societal impact of migraine and tension-type headache. Can J Neurol Sci. 1992 Aug;19(3):333-9. PMID 1393842
- [Background] Edmeads J, Findlay H, Tugwell P, Pryse-Phillips W, Nelson RF, Murray TJ. Impact of migraine and tension-type headache on life-style, consulting behaviour, and medication use: a Canadian population survey. Can J Neurol Sci. 1993 May;20(2):131-7. doi: 10.1017/s0317167100047697. PMID 8334575
- [Background] Huguet A, McGrath PJ, Stinson J, Tougas ME, Doucette S. Efficacy of psychological treatment for headaches: an overview of systematic reviews and analysis of potential modifiers of treatment efficacy. Clin J Pain. 2014 Apr;30(4):353-69. doi: 10.1097/AJP.0b013e318298dd8b. PMID 23823250